CLINICAL TRIAL: NCT01601899
Title: Molecular, Biochemical and Clinical Differences Between Stavudine and Tenofovir, Each Combined With Lamivudine and Efavirenz in South African HIV-infected Patients
Brief Title: Differences Between Stavudine and Tenofovir Each Combined With Lamivudine and Efavirenz in SA HIV-infected Patients
Acronym: CHRU01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMB decision to begin closeout process in view of April 2010 SA HAART guideline
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Colin Menezes, Consultant Infectious Diseases Physician and Lecturer, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRU01
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Mitochondrial Toxicity; Metabolic Complications
Keywords: trial; stavudine; tenofovir; mitochondria; insulin resistance; lipids; HOMA
MeSH Terms: conditions — Insulin Resistance | interventions — Stavudine; Lamivudine; efavirenz; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM A (Active Comparator): Stavudine (d4T) 30 mg po BD if wt < 60kg, or 40 mg po BD if wt > 60kg PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte
  Interventions: Drug: Stavudine
- ARM B (Active Comparator): Stavudine (d4T) 20 mg po BD if wt < 60kg, or 30 mg po BD if wt > 60kg PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte
  Interventions: Drug: Stavudine
- ARM C (Active Comparator): TDF 300 mg po QD PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Stavudine — 30 mg po BD if wt < 60kg, or 40 mg po BD if wt > 60kg
  Other Names: Lamivudine (3TC) 150mg po BD; PLUS; Efavirenz 600mg po nocte
  Arms: ARM A
Drug: Stavudine — 20 mg po BD if wt < 60kg, or 30 mg po BD if wt > 60kg
  Other Names: PLUS; Lamivudine (3TC) 150mg po BD; Efavirenz 600mg po nocte
  Arms: ARM B
Drug: Tenofovir — 300 mg po QD
  Other Names: PLUS; Lamivudine (3TC) 150mg po BD; Efavirenz 600mg po nocte
  Arms: ARM C

SUMMARY:
Even with the benefits of HIV therapy, there is a possibility that HIV-infected individuals develop metabolic complications once they initiate treatment, which may also ultimately put them at a risk for impending heart disease in the next decades.

The main mechanism through which the main HIV drugs are thought to cause these metabolic changes and organ toxicities is mitochondrial toxicity. Most of studies that have been done, have taken place in the West, but few, if any, have been done in South Africa.

The purpose of this study is to prospectively identify early changes between the two different drugs, Stavudine and Tenofovir, to assess their virological response, molecular, biochemical and clinical picture, and the possible associated change in cardiovascular risk factors, this, in the South African setting, and make recommendations to modify the current National AIDS role out programme

DETAILED DESCRIPTION:
There has been a major improvement in the survival of HIV-infected individuals with the role out highly active anti-retroviral therapy (HAART) in the public health sector by the South African Government in 2004.

Despite the unparalleled benefits of HAART, there is an increasing recognition that adverse events remain an important source of morbidity and even mortality. Knowledge of the adverse effects of different therapeutic regimes and understanding genetic factors that modulate the risk of toxicity, are important in the management of HIV/AIDS patients.

There are two regimens offered in the public sector, these contain a triple drug course, with either a nucleoside reverse transcriptase inhibitor (NRTI), a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a protease inhibitor (PI). With adherence to treatment, it is possible to convert HIV from a fatal infection to a chronic and manageable illness.

But, unfortunately, these therapeutic regimens are associated with the development of metabolic complications, such as dyslipidaemia, insulin resistance. Occasionally frank diabetes, and altered fat distribution, such as peripheral lipoatrophy and centripetal fat accumulation. There is a growing concern that these complications may lead to an increase in the long-term risk of cardiovascular disease in these individuals.

The first regime which contains stavudine, which is a NRTI. It is cheap and easy to administer in the short term but however is associated with more side effects, with relatively higher rates of long term risks of lipoatrophy, and peripheral neuropathy. It is also associated with an asymptomatic or a sometimes fatal lactic acidosis, it is also associated with complications such as myopathies and pancreatitis. However, some studies have suggested that reducing the d4T dose improves the toxicity profile while maintaining efficacy.

Tenofovir on the other hand, is a nucleotide analogue, it was approved in 2001 in the United States, and it use has grown since its approval. It is commonly used in initial therapy. It has shown to have a favourable lipid and mt DNA profile when compared to stavudine, but however it had no difference in virological response.

Clinical practice is moving increasingly towards the use of regimes that combine high levels of tolerability and efficacy. HIV-infected individuals develop a pattern similar to that of the metabolic syndrome once they initiate treatment, ultimately putting them at a risk for impending cardiovascular disease in the next decades. Most studies have been done in the West, but there is no data on patients from third world countries including South Africa.

This purpose of this study is to prospectively identify differences between the two different NRTIs, Stavudine, a nucleoside analogue (in different doses), and Tenofovir, a nucleotide analogue, to assess their virological response, molecular, biochemical and clinical pictures, and the possible associated change in cardiovascular risk factors, this, in the South African setting, and make recommendations to modify the current National AIDS role out programme

Primary Objectives

The following questions will be addressed:

1. To determine if there are any molecular differences (before and after starting treatment) between the regimens.
2. To determine the biochemical differences (before and after starting treatment) between the three regimens.
3. To determine clinical differences in patients in all three arms of treatment.

Secondary Objectives

The following questions will be addressed:

1. To determine the outcome of immune reconstitution by monitoring T-cell subsets changes.
2. To determine virological response by monitoring the viral load changes.
3. To determine which of the three treatment arms results in better adherence.
4. To determine if there are any changes in cardiovascular risk factors after treatment.

Study Design This is a randomised controlled study comparing two NRTIs, a nucleoside analogue Stavudine (standard dose, and low dose), and a nucleotide analogue Tenofovir, each combined with Lamivudine and Efavirenz in HIV-infected treatment-naïve patients to be conducted concurrently.

This study will compare the virologic response, molecular, biochemical and clinical differences between all treatment arms.

At entry, all participants will be enrolled into either Arm A, B or C after randomization.

Duration:48 weeks after randomization of the final participant.From enrollment, the participants had a minimum of four study visits.

Sample size:90 participants randomized (1:1:1) to either Arm A (30 participants), Arm B (30 participants) and Arm C (30 participants).

Population:HIV-infected, treatment-naïve patients, at least 18 years of age, with CD4+ cell count <200 cells/mm3.

At study entry, participants will be randomized (as described above) to one of the following treatment arms:

Arm A Stavudine (d4T) 30 mg po BD if wt < 60kg, or 40 mg po BD if wt > 60kg PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte

OR Arm B Stavudine (d4T) 20 mg po BD if wt < 60kg, or 30 mg po BD if wt > 60kg PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte

OR Arm C TDF 300 mg po QD PLUS Lamivudine (3TC) 150mg po BD PLUS Efavirenz 600mg po nocte

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented by a rapid HIV test or any licensed ELISA test kit, and confirmed by either a second rapid HIV test or an ELISA consistent with the Themba Lethu Clinic guidelines.
2. Age >/= 18 years,
3. CD4+ cell count < 200 cells/mm3.
4. The following laboratory values obtained within 45 days prior to study entry:

   * Absolute neutrophil count (ANC) ≥ 750/mm3
   * Hemoglobin ≥ 7.0 g/dL
   * Platelet count ≥ 50,000/mm3
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 2.5 x ULN
   * Total bilirubin ≤ 2.5 x ULN
5. Evidence of normal renal function within 45 days prior to study entry as determined by an estimated creatinine clearance of ≥60 mL/min using the Cockcroft-Gault formula:

   {[140 - age (yr)] x [weight (kg)] ÷ [72 x serum Cr (mg/dL)]} (X 0.85 in females.)
6. Participants of reproductive age (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e. who have had menses within the preceding 24 months), or who have not undergone surgical sterilization (e.g. hysterectomy, or bilateral oophorectomy or salpingotomy) must have a negative serum or urine pregnancy test within 45 days prior to study entry.
7. Participants of reproductive potential, must be willing to abstain from participation in a conception process (e.g. active attempt to become pregnant or in vitro fertilization). If participants are sexual active, that could lead to pregnancy, they must use at least one reliable form of contraception listed below while receiving protocol-specified medications and for 6 weeks after stopping the medication.

   * Male or female condoms with or without a spermicidal agent (condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission).
   * Diaphragm or cervical cap with spermicide
   * IUD
   * Hormonal-based contraception
   * Possible interactions of study drugs with estrogen-based contraceptives: LPV/RTV decrease plasma levels of ethinyl estradiol; therefore, estrogen-based contraceptives are not reliable for women receiving LPV/RTV and an alternative contraception method must be used.
   * NOTE: Participants who are not of reproductive potential (girls who have not reached menarche, women who have been post-menopausal for at least 24 consecutive months) girls and women who are not participating in sexual activity that could lead to pregnancy, or women who have undergone surgical sterilization, (e.g. hysterectomy, or bilateral oophorectomy or salpingotomy) are eligible without requiring the use of contraception.
8. Ability and willingness of participant
9. Intent to remain in current geographical area of residence for the duration of study.
10. Willingness to attend study visits as required by the study.

Exclusion Criteria:

1. Receipt of any antiretrovirals (including for purposes of occupational or sexual post exposure prophylaxis), except for SD Nevirapine taken within six months.
2. Use of systemic cancer chemotherapy, systemic investigational agents, immunomodulators (growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons) or rifampin within 30 days prior to study entry.
3. Breastfeeding or pregnancy.
4. Allergy to study drugs.
5. Any condition, including active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
6. Any serious illness requiring systemic treatment and/or hospitalization until participant either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry.
7. Involuntary incarceration in a correctional facility, for legal reasons or in a medical facility for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
changes in mitochondrial DNA copy number in adipocyte tissue | from baseline to 4 weeks
changes in gene expression in adipocyte tissue | from baseline to 4 weeks
changes in lipid levels | from baseline to 4 weeks
changes in glycaemic indices | from baseline to 4 weeks
changes in adipocytokines | from baseline to 4 weeks
changes in lipid levels | from baseline to 48 weeks
changes in glycaemic indices | from baseline to 48 weeks
changes in adipocytokines | from baseline to 48 weeks

SECONDARY OUTCOMES:
Time from randomization to virologic failure | up to 48 weeks
Time from randomization to death | up to 48 weeks
time from randomization to the first adverse event requiring discontinuation of any of the drugs that formed the initial regimen | up to 48 weeks
time from randomization to the first Grade 3 or higher adverse event. | up to 48 weeks
Time from randomization to HIV-related disease progression (defined as progression to WHO Clinical Stage 3 or 4) | up to 48 weeks
Adherence to study drug regimens as assessed by participant self-report and pill count. | up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colin N Menezes, FCP(SA), Principal Investigator — Clinical HIV Research Unit, University of the Witwatersrand; Ian Sanne, FCP(SA), Study Director — Clinical HIV Research Unit, University of the Witwatersrand
Locations (1):
- Themba Lethu Clinic, Helen Joseph Hospital, Auckland Park, Johannesburg, Gauteng, South Africa